CLINICAL TRIAL: NCT04707417
Title: Impact of Home Care for Recipients of Allogeneic Haematopoietic Stem Cell Transplantation
Brief Title: Home Care in Allogeneic Haematopoietic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anders E. L. Myhre, Consultant Haematologist, Oslo University Hospital
Other Study IDs: 212733
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Stem Cell Transplant Complications; Quality of Life; GVH - Graft Versus Host Reaction
MeSH Terms: interventions — Home Care Services

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Home care — Advanced home care

SUMMARY:
Mixed methods study with focus groups interviews and a prospective observational cohort study aimed to investigate the impact of advanced home care on transplant specific outcomes and quality of life in recipients of allogeneic hematopoietic stem cell transplantation

DETAILED DESCRIPTION:
Study of advanced home care after allogeneic haematopoietic stem cell transplantation (allo-HSCT). The main objective is to investigate the impact of home care on transplant specific variables and quality of life (QoL). The main hypothesis is that home care patients will home care patients will have significantly better measured QoL than patients receiving in-hospital care during the first 6 weeks after allo-HSCT. The study will be conducted as part of routine care at the departement of haematology, Oslo University Hospital.

There are qualitative and quantitative aspects to the study. The qualitative part involves focus groups interviews with patients that have been treated with allo-HSCT and have recieved home care and their caregivers.

In the prospective observational cohort study data will be collected to compare patients receiving home care and patients treated in-hospital (control group). Patients in both groups wil answer the questionnaire EORTC QLQ-C30 once weekly for 6 weeks. In addition transplant- and treatment-specific variables will be collected and compares between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Consent competency and written informed consent to participation
* Age ≥18
* Understanding and willing to comply with written and oral instructions in Norwegian
* Planned treatment with allo-HSCT
* ECOG performance status 0-2
* Caregiver (age ≥18) present 24 hours a day during the aplastic phase
* Travelling distance from residence to the hospital must be less than one hour.

Exclusion Criteria:

* Not meeting inclusion criteria
* Uncontrolled infection or other medical condtion unsuitable for out patient care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients planned for treatment with allogeneic stem cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
GRFS | 1 year
  GvHD-free, relapse-free survival
QoL | 6 weeks
  Quality of Life

SECONDARY OUTCOMES:
GvHD | 1 year
  Graft versus host disease
TRM | 1 year
  Transplant related mortality
Infection | 1 year
  Bacteriemia and invasive fungal disease

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Haematology, Division of Cancer Medicine, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No